CLINICAL TRIAL: NCT05276531
Title: Comparison of the Effect of Subcutaneous Progesterone and Vaginal Progesterone for Luteal Phase Support in Intrauterine Insemination
Brief Title: Comparison of the Effect of Subcutaneous Progesterone and Vaginal Progesterone for Luteal Phase Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18.10.2021-E.36477
Record Dates: First submitted 2022-03-03; First posted 2022-03-11 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Progesterone
Keywords: progesterone; iui

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- subcutaneous progesterone (Experimental): PROLUTEX® 25 mg Solution for injection, IBSA Group, Lugano, Switzerland
  Interventions: Drug: subcutaneous progesterone
- vaginal progesterone (Active Comparator): LUTINUS® 100 mg vaginal tablets, Ferring GmbH Wittland/Kiel/Germany
  Interventions: Drug: vaginal progesterone

INTERVENTIONS:
Drug: subcutaneous progesterone — clinical pregnancy rates
  Arms: subcutaneous progesterone
Drug: vaginal progesterone — clinical pregnancy rates
  Arms: vaginal progesterone

SUMMARY:
The invesigators aimed to seperate the patients,which is going to be applied IUI, to two different groups as prospective randomized controlled ;assess the efficacy of the two different way pressurised progesterone by appling intravaginal progesterone to the first group; subcutaneous to the second group.

DETAILED DESCRIPTION:
Approxymately %10-15 of the couples who are in reproductive age ,have infertility issues. %30-40 male factor ,%40-50 female factor and %20-25 both factors play a role in infertility etiology. Contributory factors of cases are %30-40 male factors, %40-50 female factors and %20-25 mixed type. Ovulation induction and intrauterine insemination(IUI) are the main treatments in infertility.IUI is accepted as the most used treatment procedure according to other assisted reproductive techniques because it has lower costs ,can be easy applied and less invasive.Luteal phase ,which is approximately 14 days,is identified as between the time of ovulation and the beginning of the menstruation period. The production of progesterone in this period,is related to the function of corpus luteum. Progesterone is used as luteal support in patients which are applied ovulation induction with gonadotropin(GND). Gonadotropin is going to be used for controlled ovarian stimulation. The treatment is going to be started on second or third day of the cycle and GND dose is going to be determined according to the patient's age, body mass index, ovary reserve and past stimulation dose answer. Treatment processed gonadotropin dose is going to be arranged according to the follicle's progress and endometrial thickness. Human chorionic gonadotropin(hCG) is going to be added to the treatment when dominant follicle's diameter reached to 17-18mm for occuring of the ovulation. Sperm obtained by density gradient method using fresh sperm 36 hours after hCG, is going to be applied to the female partner with the help of a soft catheter in the dorsalitotomy position under ultrasound guidance. The patient is going to be kept in the supine position after the procedure for 15 minutes. Each patient is going to be given a single insemination and told to resume sexual intercourse for 3 days after the procedure. Intravaginal progesterone once a day to the first group after insemination to the patients divided into two different groups with randomized controlled (LUTINUS® 100 mg vaginal tablet, Ferring GmbH Wittland/Kiel/Germany) , second group subcutaneous progesterone (PROLUTEX® 25 mg Solution for injection, IBSA Group, Lugano, Switzerland) is going to be used once a day. Clinical pregnancy rates are going to be recorded by performing a blood pregnancy test on the 15th day after the procedure. The investigators aimed to separate the patients, who are going to be applied IUI, in to two different groups as prospective randomized controlled; assess the efficacy of the two different way applied progesterone by appling intravaginal progesterone to the first group; subcutaneous to the second group.

ELIGIBILITY:
Inclusion Criteria:

* Absence of follicles larger than 10 mm on basal ultrasound
* Endometrial thickness less than 5 mm
* Patients with FSH<10 IU/ml, E2<60-80 pg/ml in the blood hormone test performed on the third day of the cycle and patients with antral follicle count above 7 on ultrasound
* Total motile sperm count greater than 10 million/ml
* 18-40 years old female, 18-50 years old male
* Anovulation, patients diagnosed with unexplained mild male factor infertility
* Female partners, who's BMI<25 kg/m²
* Being voluntarily

Exclusion Criteria:

* Other infertility reasons
* The patients who doesn't meet the criterias
* Refusing to attend to the research

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 146 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | day 15
  after iui betahcg levels blood sampling

SECONDARY OUTCOMES:
Ongoing pregnancy rate | Months 3
  Ongoing pregnancy rates 3 months after iui

CONTACTS AND LOCATIONS:
Overall Officials: Gurkan Kiran, MD, Study Chair — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erdem A, Erdem M, Atmaca S, Guler I. Impact of luteal phase support on pregnancy rates in intrauterine insemination cycles: a prospective randomized study. Fertil Steril. 2009 Jun;91(6):2508-13. doi: 10.1016/j.fertnstert.2008.04.029. Epub 2008 Aug 9. PMID 18692788
- [Background] Oktem M, Altinkaya SO, Yilmaz SA, Bozkurt N, Erdem M, Erdem A, Gumuslu S. Effect of luteal phase support after ovulation induction and intrauterine insemination. Gynecol Endocrinol. 2014;30(12):909-12. doi: 10.3109/09513590.2014.947567. Epub 2014 Aug 7. PMID 25102275
- [Background] Maher MA. Luteal phase support may improve pregnancy outcomes during intrauterine insemination cycles. Eur J Obstet Gynecol Reprod Biol. 2011 Jul;157(1):57-62. doi: 10.1016/j.ejogrb.2011.03.022. Epub 2011 Apr 21. PMID 21514032
- [Background] Ozcan P, Takmaz T. Identification of predictive factors for the probability of pregnancy following ovulation stimulation-intra-uterine insemination cycles in terms of female and male. J Obstet Gynaecol Res. 2021 Mar;47(3):893-899. doi: 10.1111/jog.14594. Epub 2021 Jan 5. PMID 33403758
- [Background] Keskin M, Aytac R. Does Luteal Phase Support Effect Pregnancy Rates in Intrauterine Insemination Cycles? A Prospective Randomised Controlled Study in a Tertiary Center. Obstet Gynecol Int. 2020 Aug 5;2020:6234070. doi: 10.1155/2020/6234070. eCollection 2020. PMID 32831851
- [Background] Khosravi D, Taheripanah R, Taheripanah A, Tarighat Monfared V, Hosseini-Zijoud SM. Comparison of oral dydrogesterone with vaginal progesteronefor luteal support in IUI cycles: a randomized clinical trial. Iran J Reprod Med. 2015 Jul;13(7):433-8. PMID 26494991
- [Background] Green KA, Zolton JR, Schermerhorn SM, Lewis TD, Healy MW, Terry N, DeCherney AH, Hill MJ. Progesterone luteal support after ovulation induction and intrauterine insemination: an updated systematic review and meta-analysis. Fertil Steril. 2017 Apr;107(4):924-933.e5. doi: 10.1016/j.fertnstert.2017.01.011. Epub 2017 Feb 24. PMID 28238492